

### Positive Parenting Program for Attention Deficit Hyperactivity Disorder: Maternal Perspective Shifts and Child Behavior Problems Reduction in a Clinical Trial

**Consent form** 

Nadia Abed Alrahman Amro

Date:30/4/2023

NCT07069621

Tel: 02-294-1999 E-Email: <u>IRB-R@aaup.edu</u> Website: www.aaup.edu

## Arab American University Institutional Review Board - Ramallah



### لجامعة العربية الأمريكية مجلس اخلاقيات البحث العلمي – رام الله

#### **INFORMED CONSENT**

رام الله – فلسطين Tel: 02-294-1999 E-Email: <u>IRB-R@aaup.edu</u> Website: www.aaup.edu

# Arab American University Institutional Review Board - Ramallah



## الجامعة العربية الأمريكية مجلس اخلاقيات البحث العلمي - رام الله

| I, |
|---|
| <u>Title of Study:</u> "Positive Parenting Program for Attention Deficit Hyperactivity Disorder: Maternal Perspective Shifts and Child Behavior Problems Reduction in a Clinical Trial" |
| Fulfillment of, degree, inPhilosophy of Nursing, in AAUP. (Name of program) |
| The nature and purpose of which has been explained to me byNadia Amro, and interpreted bynadia amro to the best of his/her ability in English. |
| I have been told about the nature of the research in terms of methodology, possible adverse effects and complications (as per Participant Information Sheet). After knowing and understanding all the possible advantages and disadvantages of this research, I voluntarily consent of my own free will to participate in the clinical research specified above. I understand that I can withdraw from this research at any time without assigning any reason whatsoever. |
| Date: Signature: (Participant) |
| IN THE PRESENCE OF: |
| Name: nadia amro |
| Designation: the researcher, nadia amro Signature: Maysa Kassabry |
| (Witness for Signature of Participant) |
| I confirm that I have explained to the patient the nature and purpose of the above-mentioned research. Date:30/4/2023 Signature: nadia amro |
| (Attending investigator) |

رام الله \_ فلسطين Tel: 02-294-1999 E-Email: <u>IRB-R@aaup.edu</u> Website: www.aaup.edu